CLINICAL TRIAL: NCT03193866
Title: COMparison Between All immunoTherapies for Multiple Sclerosis. An Observational Long-term Prospective Cohort Study of Safety, Efficacy and Patient's Satisfaction of MS Disease Modulatory Treatments in Relapsing-remitting Multiple Sclerosis
Brief Title: COMparison Between All immunoTherapies for Multiple Sclerosis.
Acronym: COMBAT-MS
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Kaiser Foundation Research Institute (Other)
Responsible Party: Principal Investigator, Fredrik Piehl, Professor, Karolinska Institutet
Other Study IDs: COMBAT-MS
Record Dates: First submitted 2017-04-20; First posted 2017-06-21 (Actual); Results first posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-03

CONDITIONS: Relapsing-remitting Multiple Sclerosis
Keywords: Immunomodulating treatment; Cohort study; Dimethyl fumarate; Fingolimod; Interferon-beta; Natalizumab; Rituximab; Glatiramer acetate
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Rituximab; Natalizumab; Fingolimod Hydrochloride; Alemtuzumab; Interferon-beta; Glatiramer Acetate; Dimethyl Fumarate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — Serum samples will be taken yearly for analysis of anti-drug antibodies. These samples will be saved in biobank.
  Additional blood samples will be taken for analyses of SARS-CoV-2 serologic response.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Rituximab — Comparisons of efficacy and safety between rituximab and all other frequently used immunomodulating drugs against multiple sclerosis
  Other Names: Natalizumab; Fingolimod; Alemtuzumab; Interferon-beta; Glatiramer acetate; Dimethyl Fumarate

SUMMARY:
The overarching goal of this study is to determine whether rituximab (RTX) offers effectiveness and safety advantages over other commonly used approved Disease-Modifying Drugs (DMT) in the largest real-world population-based structured prospective follow-up cohort of Relapsing-Remitting Multiple Sclerosis (RRMS) patients. The study will include both treatment naïve patients starting their first DMT and patients switching from a previous first line DMT (escalation/second-line).

DETAILED DESCRIPTION:
This is a prospective non-intervention observational prospective cohort study assessing the long-term safety and efficacy of RTX treatment in MS compared with other common MS DMTs regarding both clinical and radiological parameters in a real-life population of patients with MS.

A number of parameters will be assessed annually. These include baseline demographics, previous drug history and reasons for discontinuation, disability status (expanded disability status scale), relapses, safety and adverse events (AE), contrast enhancing T1 and newly appearing T2 lesions on magnetic resonance imaging, as well as a panel of patient reported outcome measures: Symbol Digit Modalities Test (SDMT); MS impact scale-29 (MSIS-29) Fatigue Scale for Motor and Cognitive Functions (FSMC), EuroQol-5 Dimensions (EQ-5D), the MS check scale and Treatment Satisfaction Questionnaire 9 (TSQM-9).

Retrospective data entered in medical charts and the Swedish MS registry will be included together with prospective annual structured follow up from inclusion into the study for a minimum of three years (three to nine years).

In a substudy - Covid Enhancement study - analyses will be performed regarding the effect of COVID-19 on people with MS as compared to non-MS individuals and also if there is any indication that a particular DMD is associated with a risk to contract a more severe COVID-19. The analyses will primarily be performed in official health care databases.

ELIGIBILITY:
INCLUSION CRITERIA:

The study population consists of all patients with Clinically Isolated Syndrome (CIS) or RRMS who;

* Initiate a first MS DMT (treatment naïve), or Initiate a second ever DMT, of a different drug class than the first, regardless of time between drugs or reason for discontinuation("switchers") from 1st Jan 2011 to 30st June 2018, and
* Are followed at any of the University clinics of Sweden, and
* Consent to participation in COMBAT-MS core, and
* Are expected to be capable to follow study assessments.

EXCLUSION CRITERIA:

- Patients with progressive forms of MS at start of therapy are not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients initiated at their first or second disease-modifying drug between January 1 2011 and June 30 2018 will be included in the trial. Up to present date, study-related data will be retrospectively controlled via individual study of patient records. Patients will be identified through the Swedish MS registry. Inclusion into the COMBAT-MS core study will be subject to written informed consent. Given the non-intervention design of the study and very limited study-specific procedures outside of clinical practise, we expect participation rates to be very high. Based on preliminary calculations from the MS registry the projected number of participants will be 3700 patients, out of which at least 1000 are treated with rituximab first or second-line.
Sampling Method: Non-Probability Sample
Enrollment: 3526 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Piehl, MD, PhD, Principal Investigator — Karolinska Institutet; Anders Svenningsson, MD, PhD, Principal Investigator — Karolinska Institutet; Anna Fogdell-Hahn, PhD, Principal Investigator — Karolinska Institutet; Ingrid Kockum, PhD, Principal Investigator — Karolinska Institutet; Thomas Frisell, PhD, Principal Investigator — Karolinska Institutet; Annette Langer-Gould, MD, PhD, Principal Investigator — Kaiser Permanent Southern California, Los Angeles, USA
Locations (1):
- Fredrik Piehl, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Note that unique patients could contribute to more than one treatment group, both with their first line and second line DMT, or exclusively in the first line or second line DMT group, as based on baseline characteristics. The 'total' automatically summed across groups should be interpreted as the total number of participants in first line DMT and second line DMT, respectively.
Units Other Than Participants: Treatment Episodes
Groups:
- RTX (First Line): Rituximab (First line)
- IFN (First Line): Interferons, first line DMT
- GA (First Line): Glatiramer acetate, first line DMT
- DMF (First Line): Dimethyl fumarate, first line DMT
- NTZ (First Line): Natalizumab, first line DMT
- RTX (Second Line): Rituximab, as first second line DMT
- DMF (Second Line): Dimethyl fumarate, as first second line DMT
- NTZ (Second Line): Natalizumab, as first second line DMT
- FGL (Second Line): Fingolimod, as first second line DMT
- TFL (Second Line): Teriflunomide, as first second line DMT
Period: First Line
Arm/Group | RTX (First Line) | IFN (First Line) | GA (First Line) | DMF (First Line) | NTZ (First Line) | RTX (Second Line) | DMF (Second Line) | NTZ (Second Line) | FGL (Second Line) | TFL (Second Line)
Started | 591; 591 Treatment Episodes | 992; 992 Treatment Episodes | 116; 116 Treatment Episodes | 416; 416 Treatment Episodes | 334; 334 Treatment Episodes | 0; 0 Treatment Episodes | 0; 0 Treatment Episodes | 0; 0 Treatment Episodes | 0; 0 Treatment Episodes | 0; 0 Treatment Episodes
Completed | 591; 591 Treatment Episodes | 992; 992 Treatment Episodes | 116; 116 Treatment Episodes | 416; 416 Treatment Episodes | 334; 334 Treatment Episodes | 0; 0 Treatment Episodes | 0; 0 Treatment Episodes | 0; 0 Treatment Episodes | 0; 0 Treatment Episodes | 0; 0 Treatment Episodes
Not Completed | 0; 0 Treatment Episodes | 0; 0 Treatment Episodes | 0; 0 Treatment Episodes | 0; 0 Treatment Episodes | 0; 0 Treatment Episodes | 0; 0 Treatment Episodes | 0; 0 Treatment Episodes | 0; 0 Treatment Episodes | 0; 0 Treatment Episodes | 0; 0 Treatment Episodes
Period: Second Line
Arm/Group | RTX (First Line) | IFN (First Line) | GA (First Line) | DMF (First Line) | NTZ (First Line) | RTX (Second Line) | DMF (Second Line) | NTZ (Second Line) | FGL (Second Line) | TFL (Second Line)
Started | 0; 0 Treatment Episodes | 0; 0 Treatment Episodes | 0; 0 Treatment Episodes | 0; 0 Treatment Episodes | 0; 0 Treatment Episodes | 748; 748 Treatment Episodes | 570; 570 Treatment Episodes | 541; 541 Treatment Episodes | 443; 443 Treatment Episodes | 161; 161 Treatment Episodes
Completed | 0; 0 Treatment Episodes | 0; 0 Treatment Episodes | 0; 0 Treatment Episodes | 0; 0 Treatment Episodes | 0; 0 Treatment Episodes | 748; 748 Treatment Episodes | 570; 570 Treatment Episodes | 541; 541 Treatment Episodes | 443; 443 Treatment Episodes | 161; 161 Treatment Episodes
Not Completed | 0; 0 Treatment Episodes | 0; 0 Treatment Episodes | 0; 0 Treatment Episodes | 0; 0 Treatment Episodes | 0; 0 Treatment Episodes | 0; 0 Treatment Episodes | 0; 0 Treatment Episodes | 0; 0 Treatment Episodes | 0; 0 Treatment Episodes | 0; 0 Treatment Episodes

BASELINE CHARACTERISTICS:
Population: Unique patients could conribute to more than one treatment group, both with their first line and second line DMT
Units Other Than Participants: Treatment Episodes
Groups:
- Total: Total of all reporting groups
Arm/Group | RTX (First Line) | IFN (First Line) | GA (First Line) | DMF (First Line) | NTZ (First Line) | RTX (Second Line) | DMF (Second Line) | NTZ (Second Line) | FGL (Second Line) | TFL (Second Line) | Total
Number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 748 | 570 | 541 | 443 | 161 | 3764
Number analyzed (Treatment Episodes) | 591 | 992 | 116 | 416 | 334 | 748 | 570 | 541 | 443 | 161 | 4912
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: First line and Second line reported in separate rows
  years
    First line: number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 0 | 0 | 0 | 0 | 0 | 2449
    First line | 36.9 (11.3) | 35.8 (10.5) | 36.9 (11.7) | 34.4 (9.7) | 31.6 (9.2) |  |  |  |  |  | 35.3 (10.6)
    Second line: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 748 | 570 | 541 | 443 | 161 | 2463
    Second line |  |  |  |  |  | 39.0 (10.5) | 40.6 (10.6) | 35.1 (9.6) | 37.3 (9.4) | 46.3 (9.8) | 38.7 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: First line and Second line reported in separate rows
  Participants
    First line: number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 0 | 0 | 0 | 0 | 0 | 2449
    First line: Female | 399 | 705 | 90 | 283 | 242 | 0 | 0 | 0 | 0 | 0 | 1719
    First line: Male | 192 | 287 | 26 | 133 | 92 | 0 | 0 | 0 | 0 | 0 | 730
    Second line: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 748 | 570 | 541 | 443 | 161 | 2463
    Second line: Female |  |  |  |  |  | 560 | 418 | 406 | 292 | 116 | 1792
    Second line: Male |  |  |  |  |  | 188 | 152 | 135 | 151 | 45 | 671
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    (all) |  |  |  |  |  |  |  |  |  |  | 0
Region of Enrollment [Number; unit: participants] — Population: First line reported separately as unique patients could contribute to more than one treatment groups, both with their first line and secoond line DMT
  participants
    number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 0 | 0 | 0 | 0 | 0 | 2449
    Sweden | 591 | 992 | 116 | 416 | 334 |  |  |  |  |  | 2449
Region of Enrollment [Number; unit: participants] — Population: Second line reported separately as unique patients could contribute to more than one treatment groups, both with their first line and secoond line DMT
  participants
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 748 | 570 | 541 | 443 | 161 | 2463
    Sweden |  |  |  |  |  | 748 | 570 | 541 | 443 | 161 | 2463
Year of DMT start [Median (Inter-Quartile Range); unit: year] — Population: First line and Second line reported in separate rows
  year
    First line: number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 0 | 0 | 0 | 0 | 0 | 2449
    First line | 2016 [2015 to 2017] | 2013 [2012 to 2014] | 2013 [2012 to 2014] | 2015 [2014 to 2017] | 2014 [2013 to 2016] |  |  |  |  |  | 2014 [2012 to 2016]
    Second line: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 748 | 570 | 541 | 443 | 161 | 2463
    Second line |  |  |  |  |  | 2016 [2014 to 2017] | 2015 [2014 to 2016] | 2013 [2012 to 2014] | 2013 [2012 to 2014] | 2015 [2015 to 2017] | 2014 [2013 to 2016]
Born in Sweden [Count of Participants; unit: Participants] — Population: First line and Second line reported in separate rows
  Participants
    First line: number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 0 | 0 | 0 | 0 | 0 | 2449
    First line | 494 | 782 | 98 | 337 | 278 |  |  |  |  |  | 1989
    Second line: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 748 | 570 | 541 | 443 | 161 | 2463
    Second line |  |  |  |  |  | 605 | 466 | 460 | 361 | 139 | 2031
Education, 12+ years [Count of Participants; unit: Participants] — n (%) with at least 12 years of education Population: First line and Second line reported in separate rows
  Participants
    First line: number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 0 | 0 | 0 | 0 | 0 | 2449
    First line | 310 | 545 | 61 | 226 | 161 |  |  |  |  |  | 1303
    Second line: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 748 | 570 | 541 | 443 | 161 | 2463
    Second line |  |  |  |  |  | 403 | 309 | 272 | 234 | 89 | 1307
Years since MS diagnosis [Mean (Standard Deviation); unit: years] — Population: First line and Second line reported in separate rows
  years
    First line: number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 0 | 0 | 0 | 0 | 0 | 2449
    First line | 1.3 (4.0) | 0.9 (3.1) | 1.7 (4.5) | 0.6 (2.3) | 0.5 (1.9) |  |  |  |  |  | 0.9 (3.2)
    Second line: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 748 | 570 | 541 | 443 | 161 | 2463
    Second line |  |  |  |  |  | 5.6 (5.5) | 7.1 (5.9) | 4.7 (4.8) | 5.6 (4.8) | 9.3 (6.9) | 6.0 (5.6)
Any relapse last year [Count of Participants; unit: Participants] — Population: First line and Second line reported in separate rows
  Participants
    First line: number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 0 | 0 | 0 | 0 | 0 | 2449
    First line | 367 | 648 | 62 | 265 | 252 |  |  |  |  |  | 1594
    Second line: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 748 | 570 | 541 | 443 | 161 | 2463
    Second line |  |  |  |  |  | 254 | 120 | 288 | 172 | 30 | 864
EDSS [Mean (Standard Deviation); unit: units on a scale] — Mean (Standard Deviation) Expanded Disability Status Scale (EDSS)
  Scale range:
  Minimum score: 0 (normal neurological examination) Maximum score: 10 (death due to multiple sclerosis)
  Lower scores indicate better outcomes (less disability). Higher scores indicate worse outcomes (more disability). Population: First line and Second line reported in separate rows
  units on a scale
    First line: number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 0 | 0 | 0 | 0 | 0 | 2449
    First line | 2.0 (1.3) | 1.6 (1.2) | 1.4 (1.2) | 1.5 (1.1) | 2.1 (1.3) |  |  |  |  |  | 1.7 (1.2)
    Second line: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 748 | 570 | 541 | 443 | 161 | 2463
    Second line |  |  |  |  |  | 2.0 (1.3) | 1.6 (1.3) | 2.2 (1.4) | 1.8 (1.3) | 1.8 (1.6) | 1.9 (1.4)
MSIS-29 physical [Mean (Standard Deviation); unit: units on a scale] — Mean (Standard Deviation) Multiple Sclerosis Impact Scale (MSIS-29) physical subscale.
  Measures patient-reported physical impact of multiple sclerosis. Scale range: Minimum score: 1 (least impact). Maximum score: 5 (highest impact). Lower scores indicate better outcomes. Higher scores indicate worse outcomes. Population: First line and Second line reported in separate rows
  units on a scale
    First line: number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 0 | 0 | 0 | 0 | 0 | 2449
    First line | 1.8 (0.8) | 1.6 (0.7) | 1.7 (0.6) | 1.7 (0.8) | 2.0 (0.9) |  |  |  |  |  | 1.8 (0.8)
    Second line: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 748 | 570 | 541 | 443 | 161 | 2463
    Second line |  |  |  |  |  | 1.7 (0.8) | 1.6 (0.7) | 1.9 (0.9) | 1.7 (0.8) | 1.7 (0.7) | 1.8 (0.8)
MSIS-29 psychological [Mean (Standard Deviation); unit: units on a scale] — Mean (Standard Deviation) Multiple Sclerosis Impact Scale (MSIS-29) psychological subscale.
  Measures patient-reported psychological impact of multiple sclerosis. Scale range: Minimum score: 1 (least impact). Maximum score: 5 (highest impact). Lower scores indicate better outcomes. Higher scores indicate worse outcomes. Population: First line and Second line reported in separate rows
  units on a scale
    First line: number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 0 | 0 | 0 | 0 | 0 | 2449
    First line | 2.4 (1.0) | 2.2 (0.9) | 2.6 (0.9) | 2.3 (1.0) | 2.6 (1.0) |  |  |  |  |  | 2.4 (1.0)
    Second line: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 748 | 570 | 541 | 443 | 161 | 2463
    Second line |  |  |  |  |  | 2.2 (1.0) | 2.0 (0.9) | 2.4 (1.0) | 2.2 (0.9) | 2.1 (1.0) | 2.2 (1.0)
Serious infection [Count of Participants; unit: Participants] — n (%) with hospitalization due to infection in the last five years Population: First line and Second line reported in separate rows
  Participants
    First line: number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 0 | 0 | 0 | 0 | 0 | 2449
    First line | 15 | 21 | 1 | 7 | 16 |  |  |  |  |  | 60
    Second line: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 748 | 570 | 541 | 443 | 161 | 2463
    Second line |  |  |  |  |  | 21 | 17 | 21 | 12 | 6 | 77
Cancer [Count of Participants; unit: Participants] — n (%) with any diagnosis of invasive cancer in the last five years Population: First line and Second line reported in separate rows
  Participants
    First line: number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 0 | 0 | 0 | 0 | 0 | 2449
    First line | 4 | 10 | 3 | 4 | 3 |  |  |  |  |  | 24
    Second line: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 748 | 570 | 541 | 443 | 161 | 2463
    Second line |  |  |  |  |  | 10 | 10 | 2 | 6 | 7 | 35
Antidepressant use [Count of Participants; unit: Participants] — n (%) with any filled prescription of antidepressant last year. Population: First line and Second line reported in separate rows
  Participants
    First line: number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 0 | 0 | 0 | 0 | 0 | 2449
    First line | 88 | 98 | 25 | 64 | 35 |  |  |  |  |  | 310
    Second line: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 748 | 570 | 541 | 443 | 161 | 2463
    Second line |  |  |  |  |  | 124 | 92 | 108 | 81 | 42 | 447
MACE [Count of Participants; unit: Participants] — n (%) with any diagnosis major adverse cardiovascular event (MACE) in the last five years Population: First line and Second line reported in separate rows
  Participants
    First line: number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 0 | 0 | 0 | 0 | 0 | 2449
    First line | 9 | 10 | 4 | 2 | 3 |  |  |  |  |  | 28
    Second line: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 748 | 570 | 541 | 443 | 161 | 2463
    Second line |  |  |  |  |  | 6 | 6 | 5 | 1 | 4 | 22
Arrhythmia [Count of Participants; unit: Participants] — n (%) with any diagnosis of arrythmia in the last five years Population: First line and Second line reported in separate rows
  Participants
    First line: number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 0 | 0 | 0 | 0 | 0 | 2449
    First line | 10 | 7 | 0 | 2 | 2 |  |  |  |  |  | 21
    Second line: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 748 | 570 | 541 | 443 | 161 | 2463
    Second line |  |  |  |  |  | 11 | 5 | 8 | 6 | 1 | 31
Diabetes [Count of Participants; unit: Participants] — n (%) with any diagnosis of diabetes in the last five years Population: First line and Second line reported in separate rows
  Participants
    First line: number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 0 | 0 | 0 | 0 | 0 | 2449
    First line | 13 | 17 | 2 | 4 | 7 |  |  |  |  |  | 43
    Second line: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 748 | 570 | 541 | 443 | 161 | 2463
    Second line |  |  |  |  |  | 17 | 12 | 6 | 5 | 2 | 42

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Disease Progression in Patients With Expanded Disability Status Scale (EDSS) <2.5 at Baseline
Description: Proportion of patients with baseline EDSS <2.5 progressing to 12 months confirmed EDSS ≥3 among those over 3 years of follow up.
  Expanded Disability Status Scale (EDSS) scale range:
  Minimum score: 0 (normal neurological examination). Maximum score: 10 (death due to multiple sclerosis) Lower scores indicate better outcomes (less disability). Higher scores indicate worse outcomes (more disability).
Time Frame: 3 years
Population: First line and Second line reported in separate rows
Measure: Count of Participants; unit: Participants
Arm/Group | RTX (First Line) | IFN (First Line) | GA (First Line) | DMF (First Line) | NTZ (First Line) | RTX (Second Line) | DMF (Second Line) | NTZ (Second Line) | FGL (Second Line) | TFL (Second Line)
Number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 748 | 570 | 541 | 443 | 161
Participants
  First line: number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 0 | 0 | 0 | 0 | 0
  First line | 20 | 50 | 5 | 14 | 7 | 0 | 0 | 0 | 0 | 0
  Second line: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 748 | 570 | 541 | 443 | 161
  Second line |  |  |  |  |  | 18 | 25 | 19 | 19 | 8
Statistical Analysis 1: Comparison: RTX (First Line) vs IFN (First Line); Data shown are adjusted difference in proportion, stratified by DMT line with rituximab as reference, from multivariable linear regression adjusted for age, sex, year of treatment start, country of birth, geographical region, education level, duration since MS diagnosis, baseline EDSS and MSIS-29 scores, history of serious infection, malignancy, major adverse cardiovascular event, arrythmia, use of antidepressants, diabetes. Confidence intervals are based on robust (Huber-White) standard errors; Test type: Superiority; Difference in proportion = 1.5, 95% CI 2-sided [-1.8 to 4.9]
Statistical Analysis 2: Comparison: RTX (First Line) vs GA (First Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = -0.2, 95% CI 2-sided [-6.8 to 6.5]
Statistical Analysis 3: Comparison: RTX (First Line) vs DMF (First Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = 1.3, 95% CI 2-sided [-1.7 to 4.3]
Statistical Analysis 4: Comparison: RTX (First Line) vs NTZ (First Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = -0.9, 95% CI 2-sided [-4.3 to 2.4]
Statistical Analysis 5: Comparison: RTX (Second Line) vs DMF (Second Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = 1.7, 95% CI 2-sided [-1.3 to 4.6]
Statistical Analysis 6: Comparison: RTX (Second Line) vs NTZ (Second Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = 0.3, 95% CI 2-sided [-2.7 to 3.3]
Statistical Analysis 7: Comparison: RTX (Second Line) vs FGL (Second Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = 1.2, 95% CI 2-sided [-2.0 to 4.4]
Statistical Analysis 8: Comparison: RTX (Second Line) vs TFL (Second Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = 2.0, 95% CI 2-sided [-3.2 to 7.1]

2. Primary Outcome: Confirmed Disease Progression in Patients With EDSS ≥2.5 at Baseline
Description: - Proportion of patients with baseline EDSS ≥2.5 experiencing 12 months confirmed EDSS increase of 1 point among those over 3 years of follow up
  Expanded Disability Status Scale (EDSS) scale range:
  Minimum score: 0 (normal neurological examination). Maximum score: 10 (death due to multiple sclerosis) Lower scores indicate better outcomes (less disability). Higher scores indicate worse outcomes (more disability).
Time Frame: 3 years
Population: First line and Second line reported in separate rows
Measure: Count of Participants; unit: Participants
Arm/Group | RTX (First Line) | IFN (First Line) | GA (First Line) | DMF (First Line) | NTZ (First Line) | RTX (Second Line) | DMF (Second Line) | NTZ (Second Line) | FGL (Second Line) | TFL (Second Line)
Number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 748 | 570 | 541 | 443 | 161
Participants
  First line: number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 0 | 0 | 0 | 0 | 0
  First line | 50 | 111 | 9 | 30 | 32 |  |  |  |  |
  Second line: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 748 | 570 | 541 | 443 | 161
  Second line |  |  |  |  |  | 50 | 57 | 47 | 37 | 9
Statistical Analysis 1: Comparison: RTX (First Line) vs IFN (First Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = 0.7, 95% CI 2-sided [-7.5 to 8.8]
Statistical Analysis 2: Comparison: RTX (First Line) vs GA (First Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = -2.9, 95% CI 2-sided [-18.5 to 12.8]
Statistical Analysis 3: Comparison: RTX (First Line) vs DMF (First Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = -0.1, 95% CI 2-sided [-8.8 to 8.6]
Statistical Analysis 4: Comparison: RTX (First Line) vs NTZ (First Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = -0.5, 95% CI 2-sided [-8.1 to 7.2]
Statistical Analysis 5: Comparison: RTX (Second Line) vs DMF (Second Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = 1.6, 95% CI 2-sided [-5.7 to 8.9]
Statistical Analysis 6: Comparison: RTX (Second Line) vs NTZ (Second Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = 1.6, 95% CI 2-sided [-4.7 to 8.0]
Statistical Analysis 7: Comparison: RTX (Second Line) vs FGL (Second Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = 0.9, 95% CI 2-sided [-6.2 to 7.9]
Statistical Analysis 8: Comparison: RTX (Second Line) vs TFL (Second Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = -1.6, 95% CI 2-sided [-10.8 to 7.5]

3. Primary Outcome: Disease-related Impact on Daily Life, Physical
Description: - Change in the MSIS-29 physical subscale (change from baseline; mean value) The Multiple Sclerosis Impact Scale (MSIS-29) physical subscale measures patient-reported physical impact of multiple sclerosis.
  Scale range: Minimum score: 1 (least impact). Maximum score: 5 (highest impact). Lower scores indicate better outcomes. Higher scores indicate worse outcomes.
Time Frame: 3 years
Population: First line and Second line reported in separate rows
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RTX (First Line) | IFN (First Line) | GA (First Line) | DMF (First Line) | NTZ (First Line) | RTX (Second Line) | DMF (Second Line) | NTZ (Second Line) | FGL (Second Line) | TFL (Second Line)
Number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 748 | 570 | 541 | 443 | 161
units on a scale
  First line: number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 0 | 0 | 0 | 0 | 0
  First line | -1.4 (16.6) | 1.1 (16.2) | -4.8 (17.7) | -1.2 (16.1) | -6.3 (18.0) |  |  |  |  |
  Second line: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 748 | 570 | 541 | 443 | 161
  Second line |  |  |  |  |  | -0.3 (14.5) | -0.5 (13.3) | -2.1 (16.4) | -1.3 (14.3) | 2.9 (16.5)
Statistical Analysis 1: Comparison: RTX (First Line) vs IFN (First Line); Data shown are adjusted mean differences, stratified by DMT line with rituximab as reference, from multivariable linear regression adjusted for age, sex, year of treatment start, country of birth, geographical region, education level, duration since MS diagnosis, baseline EDSS and MSIS-29 scores, history of serious infection, malignancy, major adverse cardiovascular event, arrhythmia, use of antidepressants, diabetes. Confidence intervals are based on robust (Huber-White) standard errors; Test type: Superiority; Mean Difference (Net) = 0.4, 95% CI 2-sided [-2.5 to 3.3]
Statistical Analysis 2: Comparison: RTX (First Line) vs GA (First Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Net) = -4.5, 95% CI 2-sided [-12.5 to 3.4]
Statistical Analysis 3: Comparison: RTX (First Line) vs DMF (First Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Net) = -0.3, 95% CI 2-sided [-2.5 to 1.8]
Statistical Analysis 4: Comparison: RTX (First Line) vs NTZ (First Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Net) = -2.5, 95% CI 2-sided [-4.9 to -0.1]
Statistical Analysis 5: Comparison: RTX (Second Line) vs DMF (Second Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Net) = -0.7, 95% CI 2-sided [-2.6 to 1.1]
Statistical Analysis 6: Comparison: RTX (Second Line) vs NTZ (Second Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Net) = -1.9, 95% CI 2-sided [-4.2 to 0.3]
Statistical Analysis 7: Comparison: RTX (Second Line) vs FGL (Second Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Net) = -1.8, 95% CI 2-sided [-4.0 to 0.3]
Statistical Analysis 8: Comparison: RTX (Second Line) vs TFL (Second Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Net) = 2.6, 95% CI 2-sided [-0.6 to 5.8]

4. Primary Outcome: Disease-related Impact on Daily Life, Psychological
Description: - Change in the MSIS-29 psychological subscale (change from baseline; mean value) The Multiple Sclerosis Impact Scale (MSIS-29) psychological subscale measures patient-reported psychological impact of multiple sclerosis.
  Scale range: Minimum score: 1 (least impact). Maximum score: 5 (highest impact). Lower scores indicate better outcomes. Higher scores indicate worse outcomes.
Time Frame: 3 years
Population: First line and Second line reported in separate rows
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RTX (First Line) | IFN (First Line) | GA (First Line) | DMF (First Line) | NTZ (First Line) | RTX (Second Line) | DMF (Second Line) | NTZ (Second Line) | FGL (Second Line) | TFL (Second Line)
Number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 748 | 570 | 541 | 443 | 161
units on a scale
  First line: number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 0 | 0 | 0 | 0 | 0
  First line | -8.5 (21.3) | -5.1 (20.7) | -23.1 (23.8) | -6.8 (20.7) | -12.2 (22.3) |  |  |  |  |
  Second line: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 748 | 570 | 541 | 443 | 161
  Second line |  |  |  |  |  | -3.7 (19.5) | -1.7 (19.3) | -6.1 (20.5) | -4.7 (19.5) | -0.3 (21.8)
Statistical Analysis 1: Comparison: RTX (First Line) vs IFN (First Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Net) = 2.3, 95% CI 2-sided [-2.2 to 6.8]
Statistical Analysis 2: Comparison: RTX (First Line) vs GA (First Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Net) = -8.3, 95% CI 2-sided [-20.3 to 3.7]
Statistical Analysis 3: Comparison: RTX (First Line) vs DMF (First Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Net) = 0.4, 95% CI 2-sided [-2.6 to 3.5]
Statistical Analysis 4: Comparison: RTX (First Line) vs NTZ (First Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Net) = -2.4, 95% CI 2-sided [-5.8 to 0.9]
Statistical Analysis 5: Comparison: RTX (Second Line) vs DMF (Second Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Net) = -0.1, 95% CI 2-sided [-2.9 to 2.7]
Statistical Analysis 6: Comparison: RTX (Second Line) vs NTZ (Second Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Net) = -1.5, 95% CI 2-sided [-4.5 to 1.6]
Statistical Analysis 7: Comparison: RTX (Second Line) vs FGL (Second Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Net) = -1.6, 95% CI 2-sided [-4.7 to 1.5]
Statistical Analysis 8: Comparison: RTX (Second Line) vs TFL (Second Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Net) = 2.3, 95% CI 2-sided [-1.7 to 6.4]

5. Secondary Outcome: Annualized Relapse Rate
Description: - Comparison of mean number of relapses per year between the different treatments
Time Frame: 3 years
Population: First line and Second line reported in separate rows
Measure: Mean (Standard Deviation); unit: percentage of relapses
Arm/Group | RTX (First Line) | IFN (First Line) | GA (First Line) | DMF (First Line) | NTZ (First Line) | RTX (Second Line) | DMF (Second Line) | NTZ (Second Line) | FGL (Second Line) | TFL (Second Line)
Number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 748 | 570 | 541 | 443 | 161
percentage of relapses
  First line: number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 0 | 0 | 0 | 0 | 0
  First line | 0.08 (0.31) | 0.59 (0.94) | 0.47 (0.73) | 0.26 (0.53) | 0.26 (0.63) |  |  |  |  |
  Second line: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 748 | 570 | 541 | 443 | 161
  Second line |  |  |  |  |  | 0.09 (0.34) | 0.22 (0.54) | 0.30 (0.67) | 0.30 (0.72) | 0.25 (0.61)
Statistical Analysis 1: Comparison: RTX (First Line) vs IFN (First Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = 0.39, 95% CI 2-sided [0.30 to 0.48]
Statistical Analysis 2: Comparison: RTX (First Line) vs GA (First Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = 0.27, 95% CI 2-sided [0.11 to 0.42]
Statistical Analysis 3: Comparison: RTX (First Line) vs DMF (First Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = 0.17, 95% CI 2-sided [0.10 to 0.23]
Statistical Analysis 4: Comparison: RTX (First Line) vs NTZ (First Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = 0.05, 95% CI 2-sided [-0.03 to 0.13]
Statistical Analysis 5: Comparison: RTX (Second Line) vs DMF (Second Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = 0.14, 95% CI 2-sided [0.08 to 0.19]
Statistical Analysis 6: Comparison: RTX (Second Line) vs NTZ (Second Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = 0.09, 95% CI 2-sided [0.01 to 0.16]
Statistical Analysis 7: Comparison: RTX (Second Line) vs FGL (Second Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = 0.14, 95% CI 2-sided [0.06 to 0.21]
Statistical Analysis 8: Comparison: RTX (Second Line) vs TFL (Second Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = 0.23, 95% CI 2-sided [0.13 to 0.33]

6. Secondary Outcome: Remaining on Drug
Description: - Proportion remaining on the index DMT after 3 years
Time Frame: 3 years
Population: First line and Second line reported in separate rows
Measure: Count of Participants; unit: Participants
Arm/Group | RTX (First Line) | IFN (First Line) | GA (First Line) | DMF (First Line) | NTZ (First Line) | RTX (Second Line) | DMF (Second Line) | NTZ (Second Line) | FGL (Second Line) | TFL (Second Line)
Number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 748 | 570 | 541 | 443 | 161
Participants
  First line: number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 0 | 0 | 0 | 0 | 0
  First line | 527 | 300 | 40 | 191 | 167 |  |  |  |  |
  Second line: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 748 | 570 | 541 | 443 | 161
  Second line |  |  |  |  |  | 662 | 307 | 299 | 260 | 76
Statistical Analysis 1: Comparison: RTX (First Line) vs IFN (First Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = -71.6, 95% CI 2-sided [-76.6 to -66.6]
Statistical Analysis 2: Comparison: RTX (First Line) vs GA (First Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = -66.3, 95% CI 2-sided [-76.3 to -56.4]
Statistical Analysis 3: Comparison: RTX (First Line) vs DMF (First Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = -47.3, 95% CI 2-sided [-53.0 to -41.7]
Statistical Analysis 4: Comparison: RTX (First Line) vs NTZ (First Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = -43.1, 95% CI 2-sided [-49.6 to -36.6]
Statistical Analysis 5: Comparison: RTX (Second Line) vs DMF (Second Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = -41.3, 95% CI 2-sided [-46.4 to -36.2]
Statistical Analysis 6: Comparison: RTX (Second Line) vs NTZ (Second Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = -33.9, 95% CI 2-sided [-39.8 to -28.0]
Statistical Analysis 7: Comparison: RTX (Second Line) vs FGL (Second Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = -33.9, 95% CI 2-sided [-39.7 to -28.0]
Statistical Analysis 8: Comparison: RTX (Second Line) vs TFL (Second Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = -49.8, 95% CI 2-sided [-58.0 to -41.6]

7. Secondary Outcome: Increase in EDSS
Description: - Comparison of yearly increase in mean EDSS between the different treatments
  Expanded Disability Status Scale (EDSS) scale range:
  Minimum score: 0 (normal neurological examination). Maximum score: 10 (death due to multiple sclerosis) Lower scores indicate better outcomes (less disability). Higher scores indicate worse outcomes (more disability).
Time Frame: 3 years
Population: First line and Second line reported in separate rows
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RTX (First Line) | IFN (First Line) | GA (First Line) | DMF (First Line) | NTZ (First Line) | RTX (Second Line) | DMF (Second Line) | NTZ (Second Line) | FGL (Second Line) | TFL (Second Line)
Number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 748 | 570 | 541 | 443 | 161
units on a scale
  First line: number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 0 | 0 | 0 | 0 | 0
  First line | -0.2 (1.2) | 0.1 (1.2) | 0.2 (1.2) | -0.2 (1.1) | -0.4 (1.2) |  |  |  |  |
  Second line: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 748 | 570 | 541 | 443 | 161
  Second line |  |  |  |  |  | -0.0 (0.9) | 0.1 (0.9) | -0.1 (1.1) | 0.1 (1.0) | 0.3 (0.9)
Statistical Analysis 1: Comparison: RTX (First Line) vs IFN (First Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.1 to 0.3]
Statistical Analysis 2: Comparison: RTX (First Line) vs GA (First Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.3 to 0.4]
Statistical Analysis 3: Comparison: RTX (First Line) vs DMF (First Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.2 to 0.1]
Statistical Analysis 4: Comparison: RTX (First Line) vs NTZ (First Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.3 to 0.1]
Statistical Analysis 5: Comparison: RTX (Second Line) vs DMF (Second Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.1 to 0.1]
Statistical Analysis 6: Comparison: RTX (Second Line) vs NTZ (Second Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.2 to 0.1]
Statistical Analysis 7: Comparison: RTX (Second Line) vs FGL (Second Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.1 to 0.2]
Statistical Analysis 8: Comparison: RTX (Second Line) vs TFL (Second Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.1 to 0.3]

8. Secondary Outcome: Proportion of Patients With at Least 1 Step Increase in EDSS
Description: - Comparison of yearly proportion of patients with at least 1 step increase in EDSS between the different treatments
  Expanded Disability Status Scale (EDSS) scale range:
  Minimum score: 0 (normal neurological examination). Maximum score: 10 (death due to multiple sclerosis) Lower scores indicate better outcomes (less disability). Higher scores indicate worse outcomes (more disability).
Time Frame: 3 years
Population: First line and Second line reported in separate rows
Measure: Count of Participants; unit: Participants
Arm/Group | RTX (First Line) | IFN (First Line) | GA (First Line) | DMF (First Line) | NTZ (First Line) | RTX (Second Line) | DMF (Second Line) | NTZ (Second Line) | FGL (Second Line) | TFL (Second Line)
Number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 748 | 570 | 541 | 443 | 161
Participants
  First line: number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 0 | 0 | 0 | 0 | 0
  First line | 108 | 272 | 43 | 83 | 44 |  |  |  |  |
  Second line: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 748 | 570 | 541 | 443 | 161
  Second line |  |  |  |  |  | 135 | 114 | 117 | 93 | 39
Statistical Analysis 1: Comparison: RTX (First Line) vs IFN (First Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = 4.8, 95% CI 2-sided [-2.2 to 11.9]
Statistical Analysis 2: Comparison: RTX (First Line) vs GA (First Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = 9.0, 95% CI 2-sided [-2.6 to 20.6]
Statistical Analysis 3: Comparison: RTX (First Line) vs DMF (First Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = -0.7, 95% CI 2-sided [-7.6 to 6.2]
Statistical Analysis 4: Comparison: RTX (First Line) vs NTZ (First Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = -2.6, 95% CI 2-sided [-9.4 to 4.1]
Statistical Analysis 5: Comparison: RTX (Second Line) vs DMF (Second Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = -2.6, 95% CI 2-sided [-8.6 to 3.4]
Statistical Analysis 6: Comparison: RTX (Second Line) vs NTZ (Second Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = 3.8, 95% CI 2-sided [-4.7 to 12.2]
Statistical Analysis 7: Comparison: RTX (Second Line) vs FGL (Second Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = 0.6, 95% CI 2-sided [-6.9 to 8.1]
Statistical Analysis 8: Comparison: RTX (Second Line) vs TFL (Second Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = 3.9, 95% CI 2-sided [-6.3 to 14.1]

9. Secondary Outcome: Proportion of Patients With No Evidence of Disease Activity (NEDA) -2
Description: - Comparison of yearly proportion of patients with No Evidence of Disease Activity (NEDA) -2 (free of exacerbations, new/enlarged T2-lesions and occurrence of CEL) between the treatments.
  Lower NEDA-2 scores indicate better outcomes. Higher NEDA-2 scores indicate worse outcomes.
Time Frame: 3 years
Population: First line and Second line reported in separate rows
Measure: Count of Participants; unit: Participants
Arm/Group | RTX (First Line) | IFN (First Line) | GA (First Line) | DMF (First Line) | NTZ (First Line) | RTX (Second Line) | DMF (Second Line) | NTZ (Second Line) | FGL (Second Line) | TFL (Second Line)
Number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 748 | 570 | 541 | 443 | 161
Participants
  First line: number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 0 | 0 | 0 | 0 | 0
  First line | 483 | 348 | 44 | 235 | 208 |  |  |  |  |
  Second line: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 748 | 570 | 541 | 443 | 161
  Second line |  |  |  |  |  | 638 | 356 | 326 | 226 | 95
Statistical Analysis 1: Comparison: RTX (First Line) vs IFN (First Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = -34.1, 95% CI 2-sided [-40.3 to -27.9]
Statistical Analysis 2: Comparison: RTX (First Line) vs GA (First Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = -32.2, 95% CI 2-sided [-43.0 to -21.5]
Statistical Analysis 3: Comparison: RTX (First Line) vs DMF (First Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = -21.8, 95% CI 2-sided [-27.9 to -15.7]
Statistical Analysis 4: Comparison: RTX (First Line) vs NTZ (First Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = -7.8, 95% CI 2-sided [-14.5 to -1.2]
Statistical Analysis 5: Comparison: RTX (Second Line) vs DMF (Second Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = -23.6, 95% CI 2-sided [-28.9 to -18.3]
Statistical Analysis 6: Comparison: RTX (Second Line) vs NTZ (Second Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = -12.7, 95% CI 2-sided [-18.9 to -6.5]
Statistical Analysis 7: Comparison: RTX (Second Line) vs FGL (Second Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = -26.5, 95% CI 2-sided [-32.8 to -20.2]
Statistical Analysis 8: Comparison: RTX (Second Line) vs TFL (Second Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = -31.7, 95% CI 2-sided [-40.1 to -23.2]

10. Secondary Outcome: Proportion of Patients With NEDA-3
Description: - Comparison of yearly proportion of patients with NEDA-3 (NEDA-2 plus no confirmed worsening of EDSS from baseline).
  Lower NEDA-3 scores indicate better outcomes. Higher NEDA-3 scores indicate worse outcomes.
Time Frame: 3 years
Population: First line and Second line reported in separate rows
Measure: Count of Participants; unit: Participants
Arm/Group | RTX (First Line) | IFN (First Line) | GA (First Line) | DMF (First Line) | NTZ (First Line) | RTX (Second Line) | DMF (Second Line) | NTZ (Second Line) | FGL (Second Line) | TFL (Second Line)
Number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 748 | 570 | 541 | 443 | 161
Participants
  First line: number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 0 | 0 | 0 | 0 | 0
  First line | 467 | 340 | 43 | 232 | 204 |  |  |  |  |
  Second line: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 748 | 570 | 541 | 443 | 161
  Second line |  |  |  |  |  | 619 | 339 | 314 | 220 | 94
Statistical Analysis 1: Comparison: RTX (First Line) vs IFN (First Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = -33.2, 95% CI 2-sided [-39.4 to -27.0]
Statistical Analysis 2: Comparison: RTX (First Line) vs GA (First Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = -30.6, 95% CI 2-sided [-41.4 to -19.8]
Statistical Analysis 3: Comparison: RTX (First Line) vs DMF (First Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = -20.8, 95% CI 2-sided [-27.0 to -14.7]
Statistical Analysis 4: Comparison: RTX (First Line) vs NTZ (First Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = -7.0, 95% CI 2-sided [-13.6 to -0.3]
Statistical Analysis 5: Comparison: RTX (Second Line) vs DMF (Second Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = -23.7, 95% CI 2-sided [-29.2 to -18.3]
Statistical Analysis 6: Comparison: RTX (Second Line) vs NTZ (Second Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = -12.3, 95% CI 2-sided [-18.6 to -6.1]
Statistical Analysis 7: Comparison: RTX (Second Line) vs FGL (Second Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = -25.3, 95% CI 2-sided [-31.7 to -19.0]
Statistical Analysis 8: Comparison: RTX (Second Line) vs TFL (Second Line); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in proportion = -29.5, 95% CI 2-sided [-38.2 to -20.8]

11. Secondary Outcome: Quality of Life Assessments
Description: Comparison of health-related quality of life measured by the European Quality of Life Five Dimensions (EQ-5D). Higher values indicate better health, and lower values indicate poorer health. The maximum theoretical value is 1. While there is no fixed minimum, scores can fall below 0, indicating health states worse than death. In this study, scores ranged from -0.59 to 1, which represent clinically relevant ranges of values.
Time Frame: 3 years
Population: First line and Second line reported in separate rows
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RTX (First Line) | IFN (First Line) | GA (First Line) | DMF (First Line) | NTZ (First Line) | RTX (Second Line) | DMF (Second Line) | NTZ (Second Line) | FGL (Second Line) | TFL (Second Line)
Number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 748 | 570 | 541 | 443 | 161
units on a scale
  First line: number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 0 | 0 | 0 | 0 | 0
  First line | 0.77 (0.24) | 0.77 (0.24) | 0.74 (0.26) | 0.81 (0.22) | 0.76 (0.26) |  |  |  |  |
  Second line: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 748 | 570 | 541 | 443 | 161
  Second line |  |  |  |  |  | 0.76 (0.24) | 0.81 (0.22) | 0.74 (0.27) | 0.79 (0.22) | 0.76 (0.24)
Statistical Analysis 1: Comparison: RTX (First Line) vs IFN (First Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.07 to 0.00]
Statistical Analysis 2: Comparison: RTX (First Line) vs GA (First Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.09 to 0.06]
Statistical Analysis 3: Comparison: RTX (First Line) vs DMF (First Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = -0.00, 95% CI 2-sided [-0.03 to 0.03]
Statistical Analysis 4: Comparison: RTX (First Line) vs NTZ (First Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.03 to 0.05]
Statistical Analysis 5: Comparison: RTX (Second Line) vs DMF (Second Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.02 to 0.04]
Statistical Analysis 6: Comparison: RTX (Second Line) vs NTZ (Second Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.01 to 0.06]
Statistical Analysis 7: Comparison: RTX (Second Line) vs FGL (Second Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [0.00 to 0.06]
Statistical Analysis 8: Comparison: RTX (Second Line) vs TFL (Second Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.06 to 0.03]

12. Secondary Outcome: Fatigue
Description: Comparison of fatigue measured by the Fatigue Scale for Motor and Cognitive Functions (FSMC).
  The fatigue scale for motor and cognitive functions (FSMC) scale range: Minimum score: 20. Maximum score: 100. Lower scores indicate better outcomes. Higher scores indicate worse outcomes.
Time Frame: 3 years
Population: First line and Second line reported in separate rows
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RTX (First Line) | IFN (First Line) | GA (First Line) | DMF (First Line) | NTZ (First Line) | RTX (Second Line) | DMF (Second Line) | NTZ (Second Line) | FGL (Second Line) | TFL (Second Line)
Number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 748 | 570 | 541 | 443 | 161
units on a scale
  First line: number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 0 | 0 | 0 | 0 | 0
  First line | 55.1 (22.9) | 52.1 (23.0) | 55.7 (22.2) | 48.3 (23.0) | 53.2 (23.2) |  |  |  |  |
  Second line: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 748 | 570 | 541 | 443 | 161
  Second line |  |  |  |  |  | 53.5 (23.0) | 49.7 (21.6) | 55.9 (23.0) | 49.3 (22.8) | 53.1 (22.7)
Statistical Analysis 1: Comparison: RTX (First Line) vs IFN (First Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [-3.3 to 5.2]
Statistical Analysis 2: Comparison: RTX (First Line) vs GA (First Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-9.4 to 6.4]
Statistical Analysis 3: Comparison: RTX (First Line) vs DMF (First Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-4.2 to 1.4]
Statistical Analysis 4: Comparison: RTX (First Line) vs NTZ (First Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = -2.6, 95% CI 2-sided [-5.9 to 0.8]
Statistical Analysis 5: Comparison: RTX (Second Line) vs DMF (Second Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-2.9 to 2.5]
Statistical Analysis 6: Comparison: RTX (Second Line) vs NTZ (Second Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-4.0 to 1.8]
Statistical Analysis 7: Comparison: RTX (Second Line) vs FGL (Second Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = -3.1, 95% CI 2-sided [-7.0 to 0.9]
Statistical Analysis 8: Comparison: RTX (Second Line) vs TFL (Second Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [-2.9 to 5.4]

13. Secondary Outcome: Treatment Satisfaction
Description: Comparison of patient satisfaction with their treatment using the Treatment Satisfaction Questionnaire (TSQ), items 1-9, restricted to patients remaining on index DMT at 3 years.
  The Treatment Satisfaction Questionnaire (TSQ), items 1-9 scale range: Minimum score: 0. Maximum score: 100. Lower scores indicate worse outcomes. Higher scores indicate better outcomes.
Time Frame: 3 years
Population: First line and Second line reported in separate rows
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RTX (First Line) | IFN (First Line) | GA (First Line) | DMF (First Line) | NTZ (First Line) | RTX (Second Line) | DMF (Second Line) | NTZ (Second Line) | FGL (Second Line) | TFL (Second Line)
Number analyzed (Participants) | 544 | 282 | 36 | 191 | 168 | 692 | 309 | 303 | 263 | 77
units on a scale
  First line: number analyzed (Participants) | 544 | 282 | 36 | 191 | 168 | 0 | 0 | 0 | 0 | 0
  First line | 50.1 (6.8) | 44.3 (7.7) | 42.8 (8.3) | 48.3 (7.1) | 49.5 (6.7) |  |  |  |  |
  Second line: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 692 | 309 | 303 | 263 | 77
  Second line |  |  |  |  |  | 49.5 (7.2) | 49.0 (6.7) | 49.5 (6.7) | 51.8 (6.3) | 51.6 (6.3)
Statistical Analysis 1: Comparison: RTX (First Line) vs IFN (First Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = -5.5, 95% CI 2-sided [-8.1 to -2.9]
Statistical Analysis 2: Comparison: RTX (First Line) vs GA (First Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = -5.9, 95% CI 2-sided [-10.9 to -1.0]
Statistical Analysis 3: Comparison: RTX (First Line) vs DMF (First Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-4.0 to -0.8]
Statistical Analysis 4: Comparison: RTX (First Line) vs NTZ (First Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-2.1 to 1.5]
Statistical Analysis 5: Comparison: RTX (Second Line) vs DMF (Second Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-2.2 to 0.6]
Statistical Analysis 6: Comparison: RTX (Second Line) vs NTZ (Second Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [-0.3 to 2.8]
Statistical Analysis 7: Comparison: RTX (Second Line) vs FGL (Second Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = 2.7, 95% CI 2-sided [0.9 to 4.6]
Statistical Analysis 8: Comparison: RTX (Second Line) vs TFL (Second Line); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = 2.1, 95% CI 2-sided [0.2 to 4.0]

14. Secondary Outcome: Rate of Serious Infections
Description: - Rate of serious infections, defined as hospitalizations where the main diagnosis included an ICD-10 diagnosis code in the national patient register in the 3 years after initiating index DMT
Time Frame: 3 years
Population: First line and Second line reported in separate rows
Measure: Number (95% Confidence Interval); unit: infections per 1000 person-years
Arm/Group | RTX (First Line) | IFN (First Line) | GA (First Line) | DMF (First Line) | NTZ (First Line) | RTX (Second Line) | DMF (Second Line) | NTZ (Second Line) | FGL (Second Line) | TFL (Second Line)
Number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 748 | 570 | 541 | 443 | 161
infections per 1000 person-years
  First line: number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 0 | 0 | 0 | 0 | 0
  First line | 12.7 [7.9 to 19.2] | 6.8 [4.2 to 10.5] | 5.8 [0.7 to 21.1] | 9.8 [5.0 to 17.1] | 12.2 [6.3 to 21.2] |  |  |  |  |
  Second line: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 748 | 570 | 541 | 443 | 161
  Second line |  |  |  |  |  | 20.2 [14.7 to 27.2] | 5.9 [2.8 to 10.9] | 6.2 [3.0 to 11.5] | 10.7 [5.9 to 18.0] | 14.9 [6.0 to 30.6]

15. Secondary Outcome: Rate of Major Adverse Cardiovascular Events (MACE)
Description: - Rate of MACE, defined as acute coronary syndrome, stroke or death from any cardiovascular cause based on corresponding ICD-codes in the national patient and cause of death registries in the 3 years after initiating index DMT
Time Frame: 3 years
Population: First line and Second line reported in separate rows
Measure: Number (95% Confidence Interval); unit: MACE per 1000 person-years
Arm/Group | RTX (First Line) | IFN (First Line) | GA (First Line) | DMF (First Line) | NTZ (First Line) | RTX (Second Line) | DMF (Second Line) | NTZ (Second Line) | FGL (Second Line) | TFL (Second Line)
Number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 748 | 570 | 541 | 443 | 161
MACE per 1000 person-years
  First line: number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 0 | 0 | 0 | 0 | 0
  First line | 1.7 [0.4 to 5.0] | 1.4 [0.4 to 3.5] | 0.0 [0.0 to 10.6] | 0.8 [0.0 to 4.5] | 0.0 [0.0 to 3.7] |  |  |  |  |
  Second line: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 748 | 570 | 541 | 443 | 161
  Second line |  |  |  |  |  | 1.3 [0.3 to 3.9] | 0.6 [0.0 to 3.3] | 1.2 [0.1 to 4.5] | 0.0 [0.0 to 2.8] | 4.2 [0.5 to 15.1]

16. Secondary Outcome: Rate of Invasive Cancer
Description: - Rate of incident invasive cancer, defined as invasive cancers based on corresponding ICD-codes in the national cancer registry in the 3 years after initiating index DMT.
Time Frame: 3 years
Population: First line and Second line reported in separate rows
Measure: Number (95% Confidence Interval); unit: invasive cancer per 1000 person-years
Arm/Group | RTX (First Line) | IFN (First Line) | GA (First Line) | DMF (First Line) | NTZ (First Line) | RTX (Second Line) | DMF (Second Line) | NTZ (Second Line) | FGL (Second Line) | TFL (Second Line)
Number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 748 | 570 | 541 | 443 | 161
invasive cancer per 1000 person-years
  First line: number analyzed (Participants) | 591 | 992 | 116 | 416 | 334 | 0 | 0 | 0 | 0 | 0
  First line | 0.6 [0.0 to 3.2] | 2.4 [1.0 to 4.9] | 2.9 [0.1 to 16.2] | 0.0 [0.0 to 3.0] | 3.0 [0.6 to 8.8] |  |  |  |  |
  Second line: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 748 | 570 | 541 | 443 | 161
  Second line |  |  |  |  |  | 1.3 [0.3 to 3.9] | 3.0 [1.0 to 6.9] | 1.2 [0.1 to 4.5] | 4.6 [1.7 to 9.9] | 0.0 [0.0 to 7.7]

ADVERSE EVENTS:
Time Frame: 4 years and 9 months, during prospective data collection between 2017 and 2022
Description: Per regulatory approval by the Swedish Medical Products Agency (MPA), the prospective data collection only included Serious Adverse Reactions (SARs) and Suspected Unexpected Serious Adverse Reactions (SUSARs), including All-Cause Mortality. Other adverse events were not collected (i.e., "0" Total Number of participants at risk). Events were collected from annual safety reports to the MPA, which did not include information on line of therapy. Thus, no stratification on therapy line was done.
Groups:
- RTX (First or Second Line): Rituximab, as first line or second line DMT
- DMF (First or Second Line): Dimethyl fumarate, as first line or second line DMT
- NTZ (First or Second Line): Natalizumab, as first line or second line DMT
- FGL (First Line): Fingolimod, first line DMT
- TFL (First Line): Teriflunomide, first line DMT
Arm/Group | RTX (First or Second Line) | IFN (First Line) | GA (First Line) | DMF (First or Second Line) | NTZ (First or Second Line) | FGL (First Line) | TFL (First Line)
All-Cause Mortality (participants affected / at risk) | 1/1184 | 0/884 | 0/97 | 0/870 | 0/767 | 0/384 | 1/138
Serious Adverse Events (participants affected / at risk) | 43/1184 | 1/884 | 0/97 | 1/870 | 3/767 | 3/384 | 3/138
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RTX (First or Second Line) (N=1184) | IFN (First Line) (N=884) | GA (First Line) (N=97) | DMF (First or Second Line) (N=870) | NTZ (First or Second Line) (N=767) | FGL (First Line) (N=384) | TFL (First Line) (N=138)
Pneumonia (Infections and infestations) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Serum sickness (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypogammaglobulinaemia (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemophilus sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervix carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abort spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corona virus infections (Infections and infestations) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lyme disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large granular lymphocytosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuroborreliosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Follicle centre lymphoma, follicular grade I, II, III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inflammatory bowel disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
COMBAT was an observational real-world study assessing the outcomes of different DMTs as used according to clinical practice. The assignment of treatments was not under investigator control, there was no randomization and no blinding of treatments. Although differences in patient characteristics at treatment start was accounted for by statistical modelling, the risk of residual confounding should be kept in mind.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-25): https://cdn.clinicaltrials.gov/large-docs/66/NCT03193866/Prot_SAP_000.pdf